CLINICAL TRIAL: NCT03273660
Title: Evaluation of the Re-volumizing Performance of Aliaxin (New Trademark)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0717
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Malar and Sub-malar Volume Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aliaxin (new trademark - IBSA Farmaceutici Italia S.r.l.) (Experimental)
  Interventions: Device: Aliaxin (new trademark - IBSA Farmaceutici Italia S.r.l.)

INTERVENTIONS:
Device: Aliaxin (new trademark - IBSA Farmaceutici Italia S.r.l.) — First treatment was performed during baseline visit, after the basal evaluations planned by the study procedure.
  0.5-1.1 ml of Aliaxin (new trademark) for emi-face was injected by needle (25-27 G) and/or cannula (25 G, 40 mm).
  A touch-up treatment (0.5-1.1 ml of Aliaxin new trademark for subject) was performed after 3-4 weeks (T1) in order to treat possible asymmetry.

SUMMARY:
Aim of the study is to evaluate the re-volumizing performance and the duration effect of the product Aliaxin (new trademark) in women aged 40-65 years with midface volume defects due to aging mechanism.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* age 40-65 years;
* FVLS 2-4;
* asking for midface volume restoration;
* available and able to return to the study site for the post-procedural follow-up examinations;
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the first aesthetic procedure) and at T1 (3-4 weeks after the first injection treatment execution, before the touch-up aestetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 6 months prior to the study start;
* performing permanent filler in the past;
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 3 months.
* dermatitis; presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy.
* anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) grade variation | Baseline (T0), 3-4 weeks after the 1st injection procedure (T1),2 months after the 1st injection procedure (T2),3 months after the 1st injection procedure (T3),6 months after the 1st injection procedure (T4),9 months after the 1st injection procedure(T5)
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  * Grade 1 (absent): no visible nasolabial fold; continuous skin line.
  * Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  * Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  * Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  * Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.
Facial Volume Loss Scale (FVLS) grade variation | Baseline (T0), 3-4 weeks after the 1st injection procedure (T1),2 months after the 1st injection procedure (T2),3 months after the 1st injection procedure (T3),6 months after the 1st injection procedure (T4),9 months after the 1st injection procedure(T5)
  Reduction of face volume loss corresponding to a decrease from the baseline of the Facial Volume Loss Scale (FVLS) where:
  * Grade 1: Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). No prominent bony landmarks. No visibility of underlying musculature.
  * Grade 2: An intermediate point between grade 1 and grade 3.
  * Grade 3: Moderate concavity of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas. Prominence of bony landmarks. May have visibility of underlying musculature.
  * Grade 4: An intermediate point between grade 3 and grade 5.
  * Grade 5: Severe indentation of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). Severe prominence of bony landmarks. Clear visibility of underlying musculature.

SECONDARY OUTCOMES:
Photographic documentation (3D pictures) | Baseline (T0), 3-4 weeks after the 1st injection procedure (T1),2 months after the 1st injection procedure (T2),3 months after the 1st injection procedure (T3),6 months after the 1st injection procedure (T4),9 months after the 1st injection procedure(T5)
  Three-dimensional pictures of the face taken by VECTRA H1 handheld imaging system.
Face volume variation | Baseline (T0), 3-4 weeks after the 1st injection procedure (T1),2 months after the 1st injection procedure (T2),3 months after the 1st injection procedure (T3),6 months after the 1st injection procedure (T4),9 months after the 1st injection procedure(T5)
  Face volume image analysis was carried on the 3D pictures taken by Vectra H1 thanks to Vectra analysis module (VAM) software

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy